CLINICAL TRIAL: NCT04451616
Title: Assessment of Progranulin and Chemokine-like Protein TAFA-5 (FAM19A5) Blood Levels in Adults With Metabolic Syndrome
Brief Title: Assessment of Progranulin and FAM19A5 Protein Blood Levels in Metabolic Syndrome
Acronym: PROG-FAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 353/20
Record Dates: First submitted 2020-06-15; First posted 2020-06-30 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Nutrition Disorders; Hypertension; Dyslipidemias; Glucose Intolerance; Glucose Metabolism Disorders; Obesity; Overweight and Obesity; Metabolic Syndrome
Keywords: Obesity; Hypertension; Dyslipidemia; Progranulin; FAM19A5; Adipokines; Metabolic syndrome
MeSH Terms: conditions — Nutrition Disorders; Hypertension; Dyslipidemias; Glucose Intolerance; Glucose Metabolism Disorders; Obesity; Overweight; Metabolic Syndrome | interventions — Blood Pressure; Pulse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Samples of blood, hair and urine will be collected. From whole-blood samples of serum and plasma will be determined. From whole-blood genetic material will be isolated. Samples of serum, plasma, whole-blood, urine and serum will be signed with patient's unique code preventing patient's data identification. Only study team will have access to samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - study group - patients with metabolic syndrome: Patients with metabolic syndrome will be included.
  Procedures:
  1. blood sample collection
  2. hair sample collection
  3. urine sample collection
  4. body composition analysis
  5. questionnaires
  6. blood pressure, pulse and blood oxygen saturation measurement
  Interventions: Diagnostic Test: Blood sample collection; Diagnostic Test: Hair sample collection; Diagnostic Test: Urine sample collection; Diagnostic Test: Body composition analysis; Diagnostic Test: Questionnaires; Diagnostic Test: Blood pressure, pulse and blood oxygen saturation measurement
- Group B - control group - patients without metabolic syndrome: Patients without metabolic syndrome will be included.
  1. blood sample collection
  2. hair sample collection
  3. urine sample collection
  4. body composition analysis
  5. questionnaires
  6. blood pressure, pulse and blood oxygen saturation measurement
  Interventions: Diagnostic Test: Blood sample collection; Diagnostic Test: Hair sample collection; Diagnostic Test: Urine sample collection; Diagnostic Test: Body composition analysis; Diagnostic Test: Questionnaires; Diagnostic Test: Blood pressure, pulse and blood oxygen saturation measurement

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Fasting blood sample will be collected from forearm vein. In the sample the concentration of: progranulin and serum FAM19A5 protein, leptin, VEGF, insulin, neopterin, adropin and selected cytokines, adipokines, myokines and chemokines, total cholesterol, low-density lipoproteins, high-density lipoproteins, triglycerides and glucose will be determined. Whole blood sample will be secured to isolate genetic material, detect and examine progranulin and FAM19A5 genes, and genes associated with the development of metabolic syndrome and with the body's mineral management. Serum mineral analysis will be performed.
Diagnostic Test: Hair sample collection — Hair sample collection will be performed. Hair mineral analysis will be performed.
Diagnostic Test: Urine sample collection — Urine sample collection will be performed. Urine mineral analysis will be performed.
Diagnostic Test: Body composition analysis — Body composition analysis with the use of electric bioimpedance will be performed.
Diagnostic Test: Questionnaires — Dietary and lifestyle interview with the use of dietary and lifestyle questionnaires and dietary diaries will be performed.
Diagnostic Test: Blood pressure, pulse and blood oxygen saturation measurement — Blood pressure, pulse and blood oxygen saturation measurements with the use of non-invasive methods will be performed.

SUMMARY:
The main objective of the study is to assess the serum levels of progranulin and FAM19A5 protein in adults with metabolic syndrome.

DETAILED DESCRIPTION:
The study is planned to be conducted on 40 adults with metabolic syndrome. As a control, it is planned to recruit 40 adults without metabolic syndrome. From all participants fasting venous blood samples, urine samples and hair samples will be collected. Next, serum progranulin and serum FAM19A5 protein concentrations will be determined in both groups. Also, serum concentration of leptin, vascular endothelial growth factor (VEGF), insulin, neopterin, adropin and selected cytokines, adipokines, myokines and chemokines, total cholesterol, low-density lipoproteins, high-density lipoproteins, triglycerides and glucose will be determined. Serum, hair and urine mineral content will be determined. In whole blood genetic analyses will be performed in order to detect and examine progranulin and FAM19A5 genes, and genes associated with the development of metabolic syndrome and genes associated with the body's mineral metabolism. Also, body composition analysis, blood pressure measurement, pulse measurement, blood oxygen saturation measurement and nutritional interview will be performed.

ELIGIBILITY:
Inclusion Criteria:

* written and informed consent of the participant to participate in the study;
* age 18-99;
* meeting at least three of the following five metabolic syndrome criteria:

  * waist circumference ≥80 cm in women and ≥94 cm in men;
  * serum triglycerides> 150 mg / dl (1.7 mmol / l) or treatment of hypertriglyceridemia;
  * HDL serum concentration <50 mg / dl (1.3 mmol / l) - in women and <40 mg / dl (1.0 mmol / l) - in men or treatment of this lipid disorder;
  * systolic blood pressure ≥ 130 mm Hg or diastolic blood pressure ≥ 85 mm Hg, or treatment of previously diagnosed hypertension;
  * fasting plasma glucose ≥100 mg / dl (5.6 mmol / l) or pharmacological treatment of type 2 diabetes.

Exclusion Criteria:

* secondary form obesity,
* substitution of progranulin or / and FAM19A5 protein,
* weight reduction above 5% of baseline body weight in the last 3 months preceding recruitment,
* liposuction and / or other fat reduction treatments,
* pacemaker, cardioverter / defibrillator,
* condition after stroke,
* Alzheimer's disease,
* fronto-temporal dementia,
* occurrence of other neurodegenerative diseases,
* occurrence of significant neurological disorders,
* occurrence of inflammatory autoimmune diseases,
* lysosomal storage diseases,
* clinically significant abnormal liver, kidney or thyroid function;
* acute or clinically significant inflammatory process in the respiratory, digestive, genitourinary tracts,
* connective tissue diseases or arthritis;
* active cancer,
* addiction to alcohol or drugs;
* pregnancy or childbirth during recruitment or 3 months before recruitment;
* current lactation or lactation within 3 months before recruitment;
* and / or any other condition which, according to researchers, would cause that participation would not be in the patient's best interest or could limit the credibility of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 people (women and men) with metabolic syndrome (study group) and 40 people (women and men) without metabolic syndrome (control group).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Progranulin | Measured at baseline
  Concentration of progranulin in serum
FAM19A5 Protein | Measured at baseline
  Concentration of FAM19A5 protein in serum

SECONDARY OUTCOMES:
Progranulin genes | Measured at baseline
  Detection and testing of progranulin genes
FAM19A5 protein genes | Measured at baseline
  Detection and testing of FAM19A5 protein genes
Leptin | Measured at baseline
  Concentration of leptin in serum
Vascular endothelial growth factor (VGEF) | Measured at baseline
  Concentration of VGEF in serum
Insulin | Measured at baseline
  Concentration of insulin in serum
Neopterin | Measured at baseline
  Concentration of neopterin in serum
Adropin | Measured at baseline
  Concentration of adropin in serum
Iron level in hair | Measured at baseline
  The content of iron will be determined in hair (atomic absorption spectrometry)
Zinc level in hair | Measured at baseline
  The content of zinc will be determined in hair (atomic absorption spectrometry)
Copper level in hair | Measured at baseline
  The content of copper will be determined in hair (atomic absorption spectrometry)
Iron level in serum | Measured at baseline
  The content of iron will be determined in serum (atomic absorption spectrometry)
Zinc level in serum | Measured at baseline
  The content of zinc will be determined in serum (atomic absorption spectrometry)
Copper level in serum | Measured at baseline
  The content of copper will be determined in serum (atomic absorption spectrometry)
Iron level in urine | Measured at baseline
  The content of iron will be determined in urine (atomic absorption spectrometry)
Zinc level in urine | Measured at baseline
  The content of zinc will be determined in urine (atomic absorption spectrometry)
Copper level in urine | Measured at baseline
  The content of copper will be determined in urine (atomic absorption spectrometry)
Body mass (BM) | Measured at baseline
  Body mass
Waist circumference (WC) | Measured at baseline
  Waist circumference
Hip circumference | Measured at baseline
  Hip circumference
Neck circumference | Measured at baseline
  Neck circumference
Body fat content | Measured at baseline
  Body fat content in bioimpedance
Muscle mass content | Measured at baseline
  Muscle mass content in bioimpedance
Total water content | Measured at baseline
  Total water content in bioimpedance
Systolic blood pressure | Measured at baseline
  Measurement of systolic blood pressure
Diastolic blood pressure | Measured at baseline
  Measurement of diastolic blood pressure
Pulse | Measured at baseline
  Measurement of pulse
Blood oxygen level | Measured at baseline
  Measurement of blood oxygen level- measured non-invasively with the use of oximeter
Total cholesterol (TCH) | Measured at baseline
  Blood concentration of total cholesterol
Low density lipoprotein (LDL) | Measured at baseline
  Blood concentration of low density lipoprotein (LDL)
High density lipoprotein (HDL) | Measured at baseline
  Blood concentration of high density lipoprotein (HDL)
Triglycerides | Measured at baseline
  Blood concentration of triglycerides
Glucose | Measured at baseline
  Blood concentration of glucose

CONTACTS AND LOCATIONS:
Overall Officials: Damian Skrypnik, MD; PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Department of Treatment of Obesity, Metabolic Disorders and Clinical Dietetics, Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No